CLINICAL TRIAL: NCT06257615
Title: The Effect of Post-discharge Education Provided Via Tele-nursing to Elderly Patients Who Had Surgery Due to Hip Fracture, on the Quality of Life and Functional Independence Levels of the Patients
Brief Title: The Effect of Post-discharge educatıon provıded vıa Tele-nursıng to Elderly patıents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HASRET YALÇINÖZ BAYSAL (Other)
Responsible Party: Sponsor-Investigator, HASRET YALÇINÖZ BAYSAL, Associate Professor, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HYALCINOZBAYSAL
Record Dates: First submitted 2023-12-22; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Tele-Nursing
Keywords: Functional Independence; Hip Fracture,; Post-Discharge Education,; Telenursing,; Quality of Life.
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients were included in the study and blinded without being informed about whether they were divided into groups or which groups they were in. Data of the research; They were coded as groups A and B by someone else under the control of the consultant researcher, who had no role in the intervention and measurements and did not know which group the patients were in, and transferred them to the SPSS program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education provided via TeleNursing (Experimental): Nursing intervention consists of 3 online video calls with educational content to the intervention group (1st, 2nd and 3rd weeks after discharge), 3 audio phone calls (4th, 5th and 6th weeks after discharge) and an educational booklet.
  Interventions: Behavioral: Education provided via TeleNursing
- Control (No Intervention): No intervention was made

INTERVENTIONS:
Behavioral: Education provided via TeleNursing — Online Video Call Online video interviews were conducted with the patients in the intervention group once in the first week (day 1-7), once in the second week (day 8-14) and once in the third week, using mobile phone programs and/or computer programs that provide video conversation opportunities. It was conducted in the form of remote online video calls, held three times in total, once within the 15-21st day.
  Voice Phone Call After audio telephone interviews and online video interviews were completed within the first three weeks after the patients in the intervention group were discharged; It was carried out using a mobile phone 3 times in total: once in the fourth week (day 22-28), once in the fifth week (day 29-35) and once in the sixth week (day 36-42).
  Other Names: Online Video Call and Voice Phone Call
  Arms: Education provided via TeleNursing

SUMMARY:
Purpose: The aim of this study is to evaluate the effect of post-discharge training given via tele-nursing to elderly patients operated for hip fracture on the quality of life and functional independence levels of the patients.

DETAILED DESCRIPTION:
Materials and Methods: This randomized controlled, pretest-posttest, single-center experimental study was conducted in a hospital between August 2022 and April 2023, with 30 patients in the intervention group and 30 patients in the control group. Nursing intervention was administered to the intervention group by three educational online video calls (1st, 2nd and 3rd weeks after discharge), three educational voice phone calls (4th, 5th and 6th weeks after discharge) and It consists of a training booklet with educational content. No intervention was applied to the control group. Research data; It was collected using the Patient Introduction Form, SF-36, FIM. Informed consent was obtained from the patients and caregivers with the permission of the ethics committee and the institution. Data analysis was done using Chi-Square, Independent T-Test and Dependent T-Test.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* Being hospitalized and operated on with a diagnosis of hip fracture as a result of a simple fall/falling from one's own level/osteoporotic fracture
* Being literate
* Not having a visual/hearing disability that would hinder communication.
* Not having a Mental Disorder (According to the statements of the patients)
* Having a primary caregiver aged 18 and over who will cooperate throughout the research,
* Having any of the available technical equipment that allows online calls (Phone, tablet, computer, etc.).

Exclusion Criteria:

* • Having previously broken a hip and been operated on

  * Being bedridden or using walking aids before the current fracture

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Quality of Life Scale | up to 7 weeks
  The scale consists of 36 items; 8 sub-dimensions as "physical function, social function, physical role limitation, emotional role limitation, mental health, vitality (energy, liveliness, vitality), pain and general health perception"; It is a multi-headed scale that includes two main dimensions: "physical and mental".Total score is not obtained from the scale. Evaluation is made based on the scores obtained separately for each subscale. The highest score that can be obtained for each question of the scale, 100, indicates good health status and increased health-related quality of life; The lowest score, 0, indicates poor health status and decreased health-related quality of life. The total score of the sub-dimensions is obtained by dividing the sum of the corresponding scores for each question of the scale items by the number of items.

SECONDARY OUTCOMES:
Functional Independence Scale | up to 7 weeks
  It determines the individual's degree of independence in physical and cognitive activities. The Functional Independence Scale consists of 18 items and measures in 2 areas: physical (motor) and cognitive.While physical function has 13 items, cognitive function domain has 5 items. Each item is evaluated between 1 and 7 points, with 1 point indicating complete dependence and 7 points indicating complete independence.

CONTACTS AND LOCATIONS:
Overall Officials: Hasret Yalcinoz Baysal, Associate Prof, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)